CLINICAL TRIAL: NCT06694818
Title: The Impact of Attentive System on Sleep Reactivity: a Study with a Participant-applied Electroencephalography in the Home Environment
Brief Title: The Impact of Attentive System on Sleep Reactivity
Acronym: SREEG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Ferini Strambi, Prof, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: in submission to CETLombardia1
Record Dates: First submitted 2024-11-11; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Insomnia Due to Anxiety and Fear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- healthy subjects not presenting insomnia symptoms (Active Comparator): Group of healthy subjects not presenting insomnia symptoms (SCI>16)
  Interventions: Behavioral: trauma film paradigm
- Group of healthy subjects presenting insomnia symptoms (Experimental): Group of healthy subjects presenting insomnia symptoms (SCI≤16)
  Interventions: Behavioral: trauma film paradigm

INTERVENTIONS:
Behavioral: trauma film paradigm — Use the trauma films as stressors to induce stress and evaluate how it affects sleep reactivity in healthy subjects with insomnia symptoms compared to healthy subjects without insomnia symptoms
  Other Names: no other intervention

SUMMARY:
Sleep Reactivity is defined as the degree to which a given amount of stress disrupts the sleep system, and it is consistent over time and across different type of stimuli. Sleep reactivity is a normal phenomenon under a certain threshold, but when it exceeds physiological threshold, this can lead to sleep disturbances that persist even following the removal of the stressor. Indeed, higher levels of sleep reactivity are associated to sleep quality depletion (i.e., increased sleep latency, reduced sleep efficiency and increased sleep fragmentation). The contribution of sleep reactivity in insomnia could be also related to altered (rapid eyes movement (REM)) REM sleep, since it plays a fundamental role in the elaboration of emotional and stressful stimuli, promoting a readjustment of the cognitive-emotional system. Hence, an alteration of REM after a stressor may prevent its proper processing and promote the disorder.

In order to, investigate this relationship this project aims to manipulate sleep reactivity to assess the differences between insomniacs and healthy controls, taking into account their attentional shifting performance and focusing on non-REM and REM sleep alterations.

DETAILED DESCRIPTION:
Among sleep disorders, insomnia is the most common, with a prevalence around 10%. It is a debilitating disorder characterized by complaints of difficulty with sleep initiation, duration, consolidation, or quality, that occurs despite adequate opportunity for sleep, and that results in daytime impairment (i.e., fatigue, daytime sleepiness, mood disorders, cognitive deficits). For the diagnosis of chronic insomnia these symptoms need to occur at least three times a week for at least three months. Its precise etiology is still unknown and widely debated. One of the most valid hypotheses proposed is the hyperarousal model of insomnia. As insomnia is the result of predisposing, precipitating factors and perpetuating factors, this model asserts that one of these factors include an increased arousal (somatic, cognitive, and cortical activation). Subjects with an altered state of arousal tend to cognitively focus on their sleep problem or general distressful events through a mechanism known as rumination. Rumination contributes to strengthen ''learned sleep preventing associations''. Therefore, in this context is important to clarify the role of stress in impacting sleep. It's known that a single stressor can elicit different reactions across individuals, and this concern the wakefulness as well as sleep. For this reason, in sleep research contexts increasing attention is given to the construct of Sleep Reactivity.

Sleep Reactivity is defined as the degree to which a given amount of stress disrupts the sleep system, and it is consistent over time and across different type of stimuli. Sleep reactivity is a normal phenomenon under a certain threshold, but when it exceeds physiological threshold, this can lead to sleep disturbances that persist even following the removal of the stressor. Indeed, higher levels of sleep reactivity are associated to sleep quality depletion (i.e., increased sleep latency, reduced sleep efficiency and increased sleep fragmentation). The contribution of sleep reactivity in insomnia could be also related to altered (rapid eyes movement (REM)) REM sleep, since it plays a fundamental role in the elaboration of emotional and stressful stimuli, promoting a readjustment of the cognitive-emotional system. Hence, an alteration of REM after a stressor may prevent its proper processing and promote the disorder.

Moreover, the AIE (Attention-Intention-Effort) pathway model describe the fundamental role of attention during the falling asleep process. According to the model, healthy sleep is an automatic and involuntary process, and it can be inhibited by selectively directing attention to it. Thus, focusing on sleep promotes the development and maintenance of insomnia. Despite that, little consideration is given to the role of attention. A better understanding of these mechanisms could aid the management of sleep reactivity by promoting attentional shifting strategies to divert focus from stressors and sleep.

In order to, investigate this relationship this project aims to manipulate sleep reactivity to assess the differences between insomniacs and healthy controls, taking into account their attentional shifting performance and focusing on non-REM and REM sleep alterations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, both male and female
* aged over 18 and under 65;
* Ability to understand and sign the informed consent

Exclusion Criteria:

* Subjects unable to read, understand, or correctly complete the procedures required by the study
* Subjects suffering from diagnosticated sleep disorders;
* Subjects suffering from substance addiction;
* Subjects who exceed the clinical cut-off for anxiety and/or depression symptoms;
* Subjects suffering from severe or degenerative neurological diseases;
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Diary | From enrollment tothe end of study at 18 days
  Participants will complete a daily Sleep Diary for 18 days, recording information each morning within 10 minutes of waking. This diary will provide data on participants' subjective sleep quality, including indicators such as perceived Sleep Efficiency (pecentual), number of awakenings, sleep latency duration (minute). These metrics will allow us to detect any changes in sleep patterns following stress induction compared to the baseline period.
Polysomnographic Recording | From enrollment to 4 days
  Using the portable Sleep Profiler device, we will capture objective data on participants' sleep in their home environment, ensuring an ecologically valid setting. This data will facilitate a comparison between two nights before and two nights after the stress intervention, examining changes in both overall sleep structure and quality and in-depth aspects of the REM phase.
  Outcomes will include: total sleep time (minutes), sleep onset latency (minutes), number of awakenings, wake after sleep onset (minutes), number of cortical arousals, percentage of specific sleep stages (stage 1, stage 2, slow wave sleep, REM sleep), number of arousal from REM sleep, EEG power, density of sleep spindles (raw number divided by the total minutes of stage 2).
Neuropsychological Attention Assessment | From enrollment to 4 days
  This assessment will include the Attention Network Test (ANT), which evaluates the three main sub-functions of attention-alerting, orienting/shifting, and executive control. Additionally, participants will complete the Stroop Task and the Go/No-Go Task to assess inhibitory control. These results will help us determine whether certain components of attention may mediate the sleep response to stress.
  Reaction times and accuracy for both tasks will be considered primary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale san Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No